CLINICAL TRIAL: NCT04174443
Title: The Efficacy and Safety of the Application of Pulsed Radiofrequency, Combined With Low-temperature Continuous Radiofrequency, to the Gasserian Ganglion for the Treatment of Primary Trigeminal Neuralgia
Brief Title: The Efficacy and Safety of Pulsed Radiofrequency Combined With Continuous Radiofrequency for the Trigeminal Neuralgia
Acronym: PRFCRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2019-266-01
Record Dates: First submitted 2019-11-17; First posted 2019-11-22 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal neuralgia; Pulsed radiofrequency; Continuous radiofrequency; High-voltage pulsed radiofrequency combined with low-temperature continuous radiofrequency
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed radiofrequency + Continuous radiofrequency (Experimental)
  Interventions: Procedure: High-voltage pulsed radiofrequency; Procedure: Low-temperature continuous radiofrequency
- Pulsed radiofrequency (Active Comparator)
  Interventions: Procedure: High-voltage pulsed radiofrequency

INTERVENTIONS:
Procedure: High-voltage pulsed radiofrequency — 2 Hz of pulsed radiofrequency will be administered at a voltage of 70 V, temperature of 42 °C, pulse width of 20 ms, and treatment time of 600 s.
Procedure: Low-temperature continuous radiofrequency — Low-temperature continuous radiofrequency will be performed at 60 °C, with a treatment time of 270 s.
  Arms: Pulsed radiofrequency + Continuous radiofrequency

SUMMARY:
Trigeminal neuralgia is a very painful condition, and radiofrequency therapy is reserved for patients who are resistant or intolerant to pharmacological therapy. Continuous radiofrequency and pulsed radiofrequency both have advantages and disadvantages. Recently, studies have found that pulsed radiofrequency combined with low-temperature (<65 °C) continuous radiofrequency increases the efficacy of the treatment, without leading to a significant increase in complications caused by nerve lesions. However, these reports have some limitations. The investigators plan to conduct a randomized, controlled study to compare the efficacy of applying high-voltage pulsed radiofrequency, with and without low-temperature continuous radiofrequency, to the gasserian ganglion for the treatment of trigeminal neuralgia. The primary outcome will be the effectiveness of the treatment after 12 months which is the percentage of participants with a modified Barrow Neurological Institute Pain Intensity Score between I-III.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with trigeminal neuralgia according to the International Classification of Headache Disorders, 3rd Edition criteria.
* Aged 18-75 years (inclusive), no sex limitation.
* Suffering from severe trigeminal neuralgia that cannot be alleviated effectively using conservative medical therapy such as carbamazepine, oxcarbazepine.
* Numeric rating scale score≥7 before the procedure.
* Agreed to sign the informed consent form.

Exclusion Criteria:

* Secondary trigeminal neuralgia such as trigeminal neuralgia attributed to a space-occupying lesion or multiple sclerosis.
* Infection at the puncture site.
* A history of psychiatric disease.
* Disorder indicated in the results of routine blood tests, hepatic function, renal function, coagulation function, electrocardiogram, or chest X-ray.
* Serious systemic diseases such as uncontrolled hypertension or diabetes, and cardiac dysfunction (II-III of the New York Heart Association classification).
* A history of abuse of narcotics.
* A history of receiving continuous radiofrequency to the gasserian ganglion or peripheral branches; glycerol rhizolysis; balloon compression; gamma knife; or any other neuroablative treatments.
* A history of receiving microvascular decompression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
The percentage of participants with a modified Barrow Neurological Institute Pain Intensity Score of I-III | Twelve months after the procedure
  The modified Barrow Neurological Institute Pain Intensity Score (I: No pain, off medications; II: Occasional pain, off medications; IIIa: No pain, continued use of medications; IIIb: Pain persists, but adequately controlled with medications; IV: Pain not adequately controlled with medications; V: No relief) will be used to evaluate the efficacy of the treatment. Twelve months after the procedure, participants with Barrow Neurological Institute scores of I-III will be defined as having received effective treatment. The primary outcome will be the effectiveness of the treatment after 12 months.

SECONDARY OUTCOMES:
The modified Barrow Neurological Institute Pain Intensity Score | On day 1; at 1 and 2 weeks; and after 1, 2, 3, 6, and 12 months following the procedure
  The modified Barrow Neurological Institute Pain Intensity Score (I: No pain, off medications; II: Occasional pain, off medications; IIIa: No pain, continued use of medications; IIIb: Pain persists, but adequately controlled with medications; IV: Pain not adequately controlled with medications; V: No relief) will be used to evaluate the efficacy of the treatment.
Numeric rating scale | On day 1; at 1 and 2 weeks; and after 1, 2, 3, 6, and 12 months following the procedure
  Pain was assessed after surgery by a numerical rating scale (0 indicates no pain, 10 indicates the most severe pain imaginable).
Dose of carbamazepine or oxcarbazepine | On day 1; at 1 and 2 weeks; and after 1, 2, 3, 6, and 12 months following the procedure
  Dose of carbamazepine or oxcarbazepine per day (mg/day)
Patient satisfaction scores on the 5-point Likert scale | After 1, 6 and 12 months following the procedure
  1: poor, 2: fair, 3: good, 4: very good, 5: excellent
The World Health Organization Quality of Life (WHOQOL)-BREF | After 1, 6 and 12 months following the procedure
  Quality of life will be measured using the World Health Organisation QoL-BREF (WHOQOL-BREF) questionnaire. The WHOQOL-BREF is a abbreviated version of the WHOQOL-100 assessment. WHOQOL-BREF is a self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall QOL and general health. Each domain's mean score can range between 4 and 20 and a higher score indicates a higher quality of life. The mean score of items within each domain is used to calculate the domain score. A transformation method converts domain scores to a 0-100 scale.
Numbness | On day 1; at 1 and 2 weeks; and after 1, 2, 3, 6, and 12 months following the procedure
  The Barrow Neurological Institute facial numbness scores (I: No facial numbness; II: Mild facial numbness, not bothersome; III: Facial Numbness, somewhat bothersome; IV: Facial numbness, very bothersome) will be used to evaluate the facial numbness.
Number of participants with anesthesia dolorosa | Within 12 months of the procedure
  The participant's facial sensation decreased, accompanied by pain
Number of participants with masticator weakness | Within 12 months of the procedure
  Occlusal dysfunction or a lower degree of masseter muscle fullness on one side when biting hard.
Number of participants with corneal anesthesia | Within 12 months of the procedure
  When touching the sclera with a cotton swab hair does not cause the eyelids to close quickly.
Number of participants with keratitis | Within 12 months of the procedure
  Eye dryness and pain, photophobia, lacrimation, excess mucus and other conditions diagnosed as keratitis by an ophthalmologist
Number of participants with adverse reactions | Within two weeks of the procedure
  Nausea, vomiting, and facial hematoma during and after the procedure; headache, dizziness, and cerebrospinal fluid leakage occurring within two weeks of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Zhao C, Ren H, Shrestha N, Meng L, Shen Y, Luo F. The efficacy of combining pulsed radiofrequency with low-temperature continuous radiofrequency for the treatment of primary trigeminal neuralgia: a randomized controlled trial. J Neurosurg. 2025 Mar 7;143(1):100-110. doi: 10.3171/2024.10.JNS241274. Print 2025 Jul 1. PMID 40053922
- [Derived] Ren H, Zhao C, Wang X, Shen Y, Meng L, Luo F. The Efficacy and Safety of the Application of Pulsed Radiofrequency, Combined With Low-Temperature Continuous Radiofrequency, to the Gasserian Ganglion for the Treatment of Primary Trigeminal Neuralgia: Study Protocol for a Prospective, Open-Label, Parall. Pain Physician. 2021 Jan;24(1):89-97. PMID 33400432